CLINICAL TRIAL: NCT04746443
Title: Impact of Covid-19 Affliction on Psychological and Mental Health of the College Students: Cross-Sectional Survey
Brief Title: Effect of Covid-19 Affliction on Psychological and Mental Health Among College Going Students: Cross-Sectional Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Snehil Dixit, Dr. Snehil Dixit, King Khalid University
Other Study IDs: ECM#2020-2501
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: college students; CORONA; COVID-19; Graduates
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STUDENTS: COLLEGE STUDENTS WITH POSITIVE COVID-19 TEST
  Interventions: Other: NOT APPLICABLE (NA)

INTERVENTIONS:
Other: NOT APPLICABLE (NA) — THE INTERVENTION GROUP IS NOT APPLICABLE TO THE CURRENT STUDY DESIGN

SUMMARY:
The study aims to study the effects of Novel corona virus (COVID-19) on the psychological and mental health of college going students. Online version of the Event Impact Scale - Revised will be used to filled by the students who got afflicted by the novel corona virus (COVID-19).

DETAILED DESCRIPTION:
Objective : To study the impact on psychological and mental health of COVID-19 affliction among college going students

Methodology:

Study Design: Cross-sectional Mode of implementation: Online surveys Population : COVID positive College students Inclusion criteria: Students positive to corona tests Exclusion criteria: students negative to corona tests

ELIGIBILITY:
Inclusion Criteria: Students positive for COVID-19 test -

Exclusion Criteria: Students negative for COVID-19 test

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: College going students
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-03-08 (Estimated); Study Completion 2021-03-08 (Estimated)

PRIMARY OUTCOMES:
EVENT IMPACT SCALE - REVISED | Within 1 month of the impact of COVID-19
  The IES-R is a 22-item self-report measure (for DSM-IV) that assesses subjective distress caused by traumatic events. It is a revised version of the older version, the 15-item IES (Horowitz, Wilner, & Alvarez, 1979). The IES-R contains seven additional items related to the hyperarousal symptoms of PTSD, which were not included in the original IES. Items correspond directly to 14 of the 17 DSM-IV symptoms of PTSD

CONTACTS AND LOCATIONS:
Overall Officials: SNEHIL DIXIT, PhD, Principal Investigator — King Khalid University
Locations (1):
- King Khalid University, Abhā, 'Asir Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The Data cannot be shared without the prior approval of the University